CLINICAL TRIAL: NCT01249716
Title: Follow-up Home Visits With Nutrition (OHE)
Brief Title: Follow-up Home Visits With Nutrition
Acronym: OHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Malnutrition
Keywords: follow-up home visit; Geriatric Disorder; rehabilitation
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: individual nutritional therapy — individual nutritional therapy provided by a registered dietician by means of three follow-up home visits

SUMMARY:
To assess the effect on geriatric patients of follow-up home visit including nutrition.

The hypothesis is that this can prevent hospital readmissions, and has a positive impact on functional abilities and quality of life

DETAILED DESCRIPTION:
Before and after the intervention the participants nutritional status, hand grip strength, functional abilities, well-being, dietary intake, level of tiredness,and activities of daily living will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients in nutritional risk

Exclusion Criteria:

* Dementia
* Expected readmissions
* Terminal disease
* Non-Danish speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
hospital readmissions | one year

SECONDARY OUTCOMES:
body weight | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Geriatric department, Herlev, Denmark

REFERENCES:
- [Background] Beck AM, Kjaer S, Hansen BS, Storm RL, Thal-Jantzen K. Study protocol: follow-up home visits with nutrition: a randomised controlled trial. BMC Geriatr. 2011 Dec 28;11:90. doi: 10.1186/1471-2318-11-90. PMID 22204420
- [Derived] Baldwin C, de van der Schueren MA, Kruizenga HM, Weekes CE. Dietary advice with or without oral nutritional supplements for disease-related malnutrition in adults. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002008. doi: 10.1002/14651858.CD002008.pub5. PMID 34931696
- [Derived] Beck AM, Kjaer S, Hansen BS, Storm RL, Thal-Jantzen K, Bitz C. Follow-up home visits with registered dietitians have a positive effect on the functional and nutritional status of geriatric medical patients after discharge: a randomized controlled trial. Clin Rehabil. 2013 Jun;27(6):483-93. doi: 10.1177/0269215512469384. Epub 2012 Dec 20. PMID 23258932